CLINICAL TRIAL: NCT00646815
Title: Insulin Sensitivity and Substrate Metabolism Before and After Treatment in Patients With Growth Hormone Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Louise Møller, Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus Sygehus, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LM2008
Record Dates: First submitted 2008-02-19; First posted 2008-03-31 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Growth Hormone Deficiency
Keywords: insulin sensitivity; substrate metabolism; fatty liver; intramyocellular lipids; growth hormone deficiency; Growth hormone deficiency (Adult)
MeSH Terms: conditions — Dwarfism, Pituitary; Insulin Resistance; Fatty Liver | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- a (Experimental): the aim of the present study is to characterize the treatment related changes in insulin sensitivity, substrate metabolism and intrahepatic-intramyocellular lipids in 12 adult patients, recently diagnosed with growth hormone deficiency
  Interventions: Drug: growth hormone (genotropin)
- Control (No Intervention): Intramyocellular, intrahepatic and intraabdominal lipid content, lean body mass and body fat percentage, are assessed in ten healthy controls matched on age, gender and BMI.

INTERVENTIONS:
Drug: growth hormone (genotropin) — Dosage regulation will follow the local recommendations of GHD treatment
  Arms: a

SUMMARY:
The purpose of this study is to further characterize the treatment related changes in insulin sensitivity, substrate metabolism and intrahepatic-intramyocellular lipids in patients with growth hormone deficiency (GHD).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Must be of legal age and competent
* Age: >18 and <60 years old
* Presently diagnosed with growth hormone deficiency; if panhypopituitary, the patient must be sufficiently substituted in the other axis´s, for at least 3 months before inclusion in the study

Exclusion Criteria:

* Alcohol consumption >21 units per week
* Malignant disease
* Pregnancy
* Magnetic implants or material in the body
* Claustrophobia
* BMI >30
* Heart disease (NYHA >2)
* Uncontrolled hypertension
* Manifest diabetes mellitus
* Change in medication, with any influence on glucose metabolism, 2 months prior to and until the end of the trial.

Controls are matched on age, gender and BMI

Inclusion Criteria:

* Written informed consent
* Must be of legal age and competent

Exclusion Criteria:

* Alcohol consumption >21 units per week
* Malignant disease
* Pregnancy
* Magnetic implants or material in the body
* Claustrophobia
* Heart disease (NYHA >2)
* Uncontrolled hypertension
* Manifest diabetes mellitus
* Change in medication, with any influence on glucose metabolism, 2 months prior to and until the end of the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity | before and after 3 months treatment with growth hormone

SECONDARY OUTCOMES:
substrate metabolism | before and after 3 months of growth hormone treatment
intrahepatic lipid content | before and after 3 months of growth hormone treatment
intramyocellular lipid content | before and after 3 months of growth hormone treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens OL Jorgensen, Professor MD, Principal Investigator — Medical Department M, Aarhus University Hospital, Aarhus, Denmark
Locations (2):
- Denmark (2):
  - Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus Sygehus, Denmark., Aarhus, Aarhus
  - Medical Department M, Aarhus University Hospital, Aarhus

REFERENCES:
- See also: Louise Møller — http://person.au.dk/da/louisem@dadlnet.dk/
- See also: Danish Data Protection Agency — http://www.datatilsynet.dk/english/